CLINICAL TRIAL: NCT00096538
Title: Pilot Study Of Valganciclovir In Patients With Classic, Non-HIV-Associated Kaposi's Sarcoma
Brief Title: Valganciclovir in Treating Patients With Classic Non-HIV-Associated Kaposi's Sarcoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); New York Presbyterian Hospital (Other); Weill Medical College of Cornell University (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-055; MSKCC-04055
Record Dates: First submitted 2004-11-09; First posted 2004-11-10 (Estimated); Results first posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-10

CONDITIONS: Sarcoma
Keywords: classic Kaposi sarcoma; recurrent Kaposi sarcoma
MeSH Terms: conditions — Sarcoma; Sarcoma, Kaposi | interventions — Valganciclovir

ARMS (1):
- valganciclovir (Experimental): Patients receive oral valganciclovir twice daily for 3 weeks and then once daily for 21 weeks in the absence of disease progression or unacceptable toxicity. All patients are followed for 1 month after completion of therapy. Patients with responding disease are followed monthly for up to 1 year.
  Interventions: Drug: valganciclovir

INTERVENTIONS:
Drug: valganciclovir

SUMMARY:
RATIONALE: Herpesvirus is found in the lesions of most patients with Kaposi's sarcoma, and may have a role in causing Kaposi's sarcoma. Valganciclovir is an antiviral drug that acts against many types of herpesviruses and may be an effective treatment for Kaposi's sarcoma.

PURPOSE: This clinical trial is studying how well valganciclovir works in treating patients with classic non-HIV-associated Kaposi's sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antitumor activity of valganciclovir in patients with classic non-HIV-associated Kaposi's sarcoma (KS).

Secondary

* Determine the effect of this drug on lytic and latent human herpesvirus-8 gene expression in KS lesions of these patients.
* Determine the effect of this drug on the markers of angiogenesis in KS lesions of these patients.
* Determine the safety and tolerability of this drug in these patients.

OUTLINE: This is a pilot study.

Patients receive oral valganciclovir twice daily for 3 weeks and then once daily for 21 weeks in the absence of disease progression or unacceptable toxicity.

All patients are followed for 1 month after completion of therapy. Patients with responding disease are followed monthly for up to 1 year.

PROJECTED ACCRUAL: A total of 15 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed classic Kaposi's sarcoma (KS) involving the skin

  * Non-HIV-associated disease

    * HIV negative
* Measurable disease

  * At least 8 KS lesions with ≥ 5 marker lesions measurable in 2 dimensions AND ≥ 3 other lesions measuring ≥ 1 cm in diameter

    * Two 3 mm punch biopsies of a non-marker lesion entirely composed of KS
  * Irradiated cutaneous lesions may not be used as indicator lesions
* No known active visceral KS or symptomatic KS-related edema that would preclude function or require cytotoxic chemotherapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* At least 12 months

Hematopoietic

* Hemoglobin ≥ 8 g/dL
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 3 times ULN

Renal

* Creatinine clearance ≥ 50 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after study participation
* No hypersensitivity to valganciclovir or ganciclovir
* No other neoplasia requiring cytotoxic therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior biological therapy for KS
* No concurrent immunotherapy

Chemotherapy

* More than 4 weeks since prior chemotherapy for KS
* No concurrent chemotherapy

Endocrine therapy

* No concurrent corticosteroid treatment except for replacement doses (equivalent to 20 mg of hydrocortisone per day)

Radiotherapy

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy for KS
* No concurrent radiotherapy

Surgery

* Not specified

Other

* More than 14 days since prior acute treatment for infection (other than oral thrush or genital herpes) or other serious medical illness
* More than 60 days since prior local therapy for any KS indicator lesion unless the lesion showed documented progression since treatment
* More than 4 weeks since prior local therapy for KS
* More than 4 weeks since prior investigational agents
* More than 4 weeks since other prior antineoplastic therapy for KS
* No other concurrent antiviral therapy
* No other concurrent investigational agents
* No other concurrent systemic therapy for KS

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2004-04; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan E. Krown, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan - Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Valganciclovir
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Valganciclovir
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate Every 4 Weeks
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Valganciclovir
Number analyzed (Participants) | 5
participants
  Progression of Disease | 4
  Stable Disease | 1

ADVERSE EVENTS:
Arm/Group | Valganciclovir
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valganciclovir (N=6)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valganciclovir (N=6)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (6)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes